CLINICAL TRIAL: NCT02856984
Title: International Prospective Observational Cohort Study of Zika in Infants
Brief Title: Zika in Infants and Pregnancy (ZIP)
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GN ZIKA
Record Dates: First submitted 2016-07-20; First posted 2016-08-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Zika Virus Disease (Disorder)
Keywords: Pregnancy; Infant
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal samples from urine, blood, genital secretions, saliva, and breast milk, and when available amniotic fluid and tissue; infant urine, blood, and saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ZIKV infected women: The study will prospectively enroll pregnant women up to 17 weeks and 6 days gestation and follow them through their pregnancy for clinical evidence of acute ZIKV infection while controlling for potential confounders. All pregnant women will be followed throughout the pregnancy, delivery, and 6 weeks postpartum. Outcomes in women, the developing fetus, and infants will be assessed.
- Control (uninfected women): The women who remain uninfected will serve as the internal comparison group. The infants who remain uninfected at delivery and throughout the follow-up period will serve as the internal comparison group.

SUMMARY:
The overall objective of this multisite, multicountry Zika in Infants and Pregnancy (ZIP) study is to assess the strength of the association between Zika virus infection (ZIKV) during pregnancy and adverse maternal/fetal outcomes and the risk of vertical transmission. The study will prospectively enroll a cohort of pregnant women up to 17 weeks and 6 days gestation and subjects at any gestational age with acute Zika infection, confirmed by serology or PCR (polymerase chain reaction) test. The study will follow these women through their pregnancy to identify for clinical evidence of acute ZIKV, while controlling for potential confounders. Outcomes in the women, the developing fetus, and infants will be assessed. All protocol-specified data will be recorded and entered in a central data management system for the purposes of analysis of composite data from the study.

DETAILED DESCRIPTION:
The overall objective of this multisite, multicountry Zika in Infants and Pregnancy (ZIP) study is to assess the strength of the association between Zika virus infection (ZIKV) during pregnancy and adverse maternal/fetal outcomes and the risk of vertical transmission. The study will prospectively enroll a cohort of pregnant women up to 17 weeks and 6 days gestation and subjects at any gestational age with acute Zika infection, confirmed by serology or PCR (polymerase chain reaction) test. The study will follow these women through their pregnancy to identify for clinical evidence of acute ZIKV, while controlling for potential confounders. Outcomes in the women, the developing fetus, and infants will be assessed. All protocol-specified data will be recorded and entered in a central data management system for the purposes of analysis of composite data from the study.

The study will recruit up to10,000 pregnant women in their first trimester from ZIKV-endemic regions and follow them longitudinally to study the impact of incident ZIKV during pregnancy on maternal, fetal, and newborn outcomes. Researchers will identify cases of incident ZIKV among pregnant women by monitoring for symptoms of Zika-like illness and performing serial laboratory sampling for diagnosis of seroconversion and viral shedding. After delivery, infants born with evidence of ZIKV or born to mothers diagnosed with incident virus infection will be followed in a prospective longitudinal cohort for at least 1 year. In addition, a control group of infants born to mothers without evidence of ZIKV during pregnancy will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >15 years
* Assent and consent as required per local country regulations
* Confirmation of pregnancy by beta human chorionic gonadotropin (hCG) measurement in blood/urine or ultrasound confirmation of pregnancy with fetal heart tones present
* Pregnant women up to 17 weeks and 6 days gestation and subjects at any gestational age with acute Zika infection, confirmed by serology or PCR (polymerase chain reaction) test.

Exclusion Criteria: Pregnant Women

* Women who cannot adhere to proposed testing schedule
* Pregnant women enrolled in other research including other ZIKV research

Inclusion Criteria (newborn)

* All infants born to women enrolled in the observational cohort are eligible for enrollment

Exclusion Criteria (newborn)

* Mother or custodial parent does not consent to have child participate
* Infants born to mothers that are not part of the ZIP cohort study

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit up to 10,000 pregnant women up to 17 weeks and 6 days gestation and subjects at any gestational age with acute Zika infection, confirmed by serology or PCR (polymerase chain reaction) test from ZIKV-endemic regions and follow them longitudinally to study the impact of incident ZIKV during pregnancy on maternal, fetal, and newborn outcomes. Researchers will identify cases of incident ZIKV among pregnant women by monitoring for symptoms of Zika-like illness and performing serial laboratory sampling for diagnosis of seroconversion and viral shedding. After delivery, infants born with evidence of ZIKV or born to mothers diagnosed with incident virus infection will be followed in a prospective longitudinal cohort for at least 1 year. In addition, a control group of infants born to mothers without evidence of ZIKV during pregnancy will be followed.
Sampling Method: Probability Sample
Enrollment: 6461 (Actual)
Dates: Start 2016-06; Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Incidence of congenital malformations for ZIKV infected participants | Time of birth of infant
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV infected participants | 3 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV infected participants | 6 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV infected participants | 12 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV infected participants | Time of birth of infant
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, central nervous system (CNS) malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV infected participants | 3 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, central nervous system (CNS) malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV infected participants | 6 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, central nervous system (CNS) malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV infected participants | 12 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, central nervous system (CNS) malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of congenital malformations for ZIKV symptomatic participants | Time of birth of infant
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV symptomatic participants | 3 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV symptomatic participants | 6 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of congenital malformations for ZIKV symptomatic participants | 12 months of age
  To measure the incidence of congenital malformations in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV symptomatic participants | Time of birth of infant
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, CNS malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV symptomatic participants | 3 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, CNS malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV symptomatic participants | 6 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, CNS malformations, hydrops, and ocular abnormalities) in fetuses/infants.
Incidence of adverse fetal outcomes for ZIKV symptomatic participants | 12 months of age
  To measure the incidence of adverse fetal outcomes (including microcephaly, fetal demise, neonatal death, CNS malformations, hydrops, and ocular abnormalities) in fetuses/infants.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ximenes, MD, Principal Investigator — Departamento de Medicina Tropical da Universidade Federal de Pernambuco-UFPE; William Britt, MD, Principal Investigator — University of Alabama Birmingham School of Medicine; Marisa Mussi, MD, Principal Investigator — Ribeirão Preto Medical School, University of São Paulo; Albert Ko, MD, Principal Investigator — Yale University, Laboratory of Epidemiology and Public Health; Deolinda Scalabrin, Principal Investigator — Centro de Pesquisas Gonçalo Moniz, Fundação Oswaldo Cruz/MS; Marisa Elisabeth Lopes, Principal Investigator — Instituto Fernandes Figueira - FIOCRUZ; Ana Garces, MD, Principal Investigator — Fundación para la Alimentación y Nutrición de Centro América y Panamá (INCAP); Jose Cordero, MD, Principal Investigator — University of Georgia; Carmen Milagros Velez Vega, PhD, Principal Investigator — University of Puerto Rico; George Seage, MD, Principal Investigator — Harvard University School of Public Health; Carmen Zorilla, MD, Principal Investigator — University of Puerto Rico; Eva Harris, PhD, Principal Investigator — University of Californina Berkeley; Angel Balmaseda, Principal Investigator — MINSA Central; Juan F Arias, MD, Principal Investigator — St. Jude Children's Research Hospital; Jill Lebov, PhD, Principal Investigator — RTI International; Teresa Ochoa Woodell, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (10):
- Brazil (4):
  - Centro de Pesquisas Gonçalo Moniz, Fundação Oswaldo Cruz/MS; Rue Waldemar Falcao, Salvador, Estado de Bahia
  - Departamento de Medicina Tropical da Universidade Federal de Pernambuco-UFPE, Recife, Pernambuco
  - Instituto Fernandes Figueira - FIOCRUZ, Rio de Janeiro, Rio de Janeiro
  - Ribeirão Preto Medical School, University of São Paulo, Av. Bandeirantes, 3900 - Monte Alegre, Ribeirão Preto, São Paulo
- Centro Medico Imbanaco, Cali, Colombia
- Fundación para la Alimentación y Nutrición de Centro América y Panamá (INCAP), Guatemala City, Guatemala
- MINSA Central, Managua, Nicaragua
- Universidad Peruana, Lima, Peru
- Puerto Rico (2):
  - University of Puerto Rico Medical Sciences Campus, San Juan
  - University of Puerto Rico - Recinto de Río Piedras, San Juan

IPD SHARING:
Plan to Share IPD: Yes
de-identified participant data will be entered into the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (N-DASH) system.
Time Frame: IPD Sharing Time Frame: March 2022

REFERENCES:
- [Background] WHO statement on the first meeting of the International Health Regulations (2005) (IHR 2005) Emergency Committee on Zika virus and observed increase in neurological disorders and neonatal malformations; 1 February 2016. Available at http://www.who.int/ mediacentre/news/statements/2016/1st-emergency-committee-zika/en/
- [Background] Petersen EE, Staples JE, Meaney-Delman D, Fischer M, Ellington SR, Callaghan WM, Jamieson DJ. Interim Guidelines for Pregnant Women During a Zika Virus Outbreak--United States, 2016. MMWR Morb Mortal Wkly Rep. 2016 Jan 22;65(2):30-3. doi: 10.15585/mmwr.mm6502e1. PMID 26796813
- [Background] Powles R, Smith C, Milan S, Treleaven J, Millar J, McElwain T, Gordon-Smith E, Milliken S, Tiley C. Human recombinant GM-CSF in allogeneic bone-marrow transplantation for leukaemia: double-blind, placebo-controlled trial. Lancet. 1990 Dec 8;336(8728):1417-20. doi: 10.1016/0140-6736(90)93111-2. PMID 1978880
- [Background] CDC. Chikungunya virus. Atlanta, GA: US Department of Health and Human Services, CDC; 2015. http://www.cdc.gov/chikungunya/hc/clinicalevaluation.html
- [Background] Dengue: Guidelines for Diagnosis, Treatment, Prevention and Control: New Edition. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK143157/ PMID 23762963
- [Background] CDC Zika Virus; Areas with Zika http://www.cdc.gov/zika/geo/index.html
- [Background] Oliveira Melo AS, Malinger G, Ximenes R, Szejnfeld PO, Alves Sampaio S, Bispo de Filippis AM. Zika virus intrauterine infection causes fetal brain abnormality and microcephaly: tip of the iceberg? Ultrasound Obstet Gynecol. 2016 Jan;47(1):6-7. doi: 10.1002/uog.15831. No abstract available. PMID 26731034
- [Background] CDC. West Nile virus: insect repellent use & safety. Atlanta, GA: US Department of Health and Human Services, CDC; 2015. http://www.cdc.gov/westnile/faq/repellent.html.
- [Background] CDC. Zika virus. Atlanta, GA: US Department of Health and Human Services, CDC; 2015. http://www.cdc.gov/zika/index.html
- [Background] Oduyebo T, Petersen EE, Rasmussen SA, Mead PS, Meaney-Delman D, Renquist CM, Ellington SR, Fischer M, Staples JE, Powers AM, Villanueva J, Galang RR, Dieke A, Munoz JL, Honein MA, Jamieson DJ. Update: Interim Guidelines for Health Care Providers Caring for Pregnant Women and Women of Reproductive Age with Possible Zika Virus Exposure - United States, 2016. MMWR Morb Mortal Wkly Rep. 2016 Feb 12;65(5):122-7. doi: 10.15585/mmwr.mm6505e2. PMID 26866840
- [Background] Babaliche P, Doshi D. Catching Dengue Early: Clinical Features and Laboratory Markers of Dengue Virus Infection. J Assoc Physicians India. 2015 May;63(5):38-41. PMID 26591143
- [Background] Wahala WM, Silva AM. The human antibody response to dengue virus infection. Viruses. 2011 Dec;3(12):2374-95. doi: 10.3390/v3122374. Epub 2011 Nov 25. PMID 22355444
- [Background] Gibney KB, Edupuganti S, Panella AJ, Kosoy OI, Delorey MJ, Lanciotti RS, Mulligan MJ, Fischer M, Staples JE. Detection of anti-yellow fever virus immunoglobulin m antibodies at 3-4 years following yellow fever vaccination. Am J Trop Med Hyg. 2012 Dec;87(6):1112-5. doi: 10.4269/ajtmh.2012.12-0182. Epub 2012 Oct 29. PMID 23109371
- [Background] Roehrig JT, Nash D, Maldin B, Labowitz A, Martin DA, Lanciotti RS, Campbell GL. Persistence of virus-reactive serum immunoglobulin m antibody in confirmed west nile virus encephalitis cases. Emerg Infect Dis. 2003 Mar;9(3):376-9. doi: 10.3201/eid0903.020531. PMID 12643836
- [Background] http://www.salud.gov.pr/Estadisticas-Registros-y-Publicaciones/Informes %20Arbovirales/Reporte%20ArboV%20semana%204-2016.pdf
- [Background] Chervenak FA, Jeanty P, Cantraine F, Chitkara U, Venus I, Berkowitz RL, Hobbins JC. The diagnosis of fetal microcephaly. Am J Obstet Gynecol. 1984 Jul 1;149(5):512-7. doi: 10.1016/0002-9378(84)90027-9. PMID 6742021
- [Background] Chervenak FA, Rosenberg J, Brightman RC, Chitkara U, Jeanty P. A prospective study of the accuracy of ultrasound in predicting fetal microcephaly. Obstet Gynecol. 1987 Jun;69(6):908-10. PMID 3554067
- [Background] Kurtz AB, Wapner RJ, Rubin CS, Cole-Beuglet C, Ross RD, Goldberg BB. Ultrasound criteria for in utero diagnosis of microcephaly. J Clin Ultrasound. 1980 Feb;8(1):11-6. doi: 10.1002/jcu.1870080104. PMID 6766470
- [Background] Hutchon DJ. Fetal ultrasound biometry: 1. Head reference values. Br J Obstet Gynaecol. 1999 Aug;106(8):875-6. doi: 10.1111/j.1471-0528.1999.tb08417.x. No abstract available. PMID 10453845
- [Background] Berger I. Prenatal microcephaly: can we be more accurate? J Child Neurol. 2009 Jan;24(1):97-100. doi: 10.1177/0883073808321045. PMID 19168823
- [Background] Julie A Boom; Microcephaly in infants and children: Etiology and evaluation UpToDate http://www.uptodate.com/contents/microcephaly-in-infants-and-children- etiology-and-evaluation?source=machineLearning&search=microcephaly+in +pregnacy&selectedTitle=2~130§ionRank=3&anchor=H55603463#H55603463 Accessed on February 16, 2016
- [Background] Tolmie JL, McNay M, Stephenson JB, Doyle D, Connor JM. Microcephaly: genetic counselling and antenatal diagnosis after the birth of an affected child. Am J Med Genet. 1987 Jul;27(3):583-94. doi: 10.1002/ajmg.1320270311. PMID 3307411
- [Background] Atkinson B, Hearn P, Afrough B, Lumley S, Carter D, Aarons EJ, Simpson AJ, Brooks TJ, Hewson R. Detection of Zika Virus in Semen. Emerg Infect Dis. 2016 May;22(5):940. doi: 10.3201/eid2205.160107. No abstract available. PMID 27088817
- [Background] Medscape Medical News; FDA Issues Guidance to Protect Blood Supply From Zika Virus http://www.medscape.com/viewarticle/858976? nlid=100283_3901&src=wnl_newsalrt_160216_MSCPEDIT&uac=17333MK&impID=993653&faf=1
- [Background] Sarno M, Sacramento GA, Khouri R, do Rosario MS, Costa F, Archanjo G, Santos LA, Nery N Jr, Vasilakis N, Ko AI, de Almeida AR. Zika Virus Infection and Stillbirths: A Case of Hydrops Fetalis, Hydranencephaly and Fetal Demise. PLoS Negl Trop Dis. 2016 Feb 25;10(2):e0004517. doi: 10.1371/journal.pntd.0004517. eCollection 2016 Feb. PMID 26914330
- [Background] Brasil P, Pereira JP Jr, Moreira ME, Ribeiro Nogueira RM, Damasceno L, Wakimoto M, Rabello RS, Valderramos SG, Halai UA, Salles TS, Zin AA, Horovitz D, Daltro P, Boechat M, Raja Gabaglia C, Carvalho de Sequeira P, Pilotto JH, Medialdea-Carrera R, Cotrim da Cunha D, Abreu de Carvalho LM, Pone M, Machado Siqueira A, Calvet GA, Rodrigues Baiao AE, Neves ES, Nassar de Carvalho PR, Hasue RH, Marschik PB, Einspieler C, Janzen C, Cherry JD, Bispo de Filippis AM, Nielsen-Saines K. Zika Virus Infection in Pregnant Women in Rio de Janeiro. N Engl J Med. 2016 Dec 15;375(24):2321-2334. doi: 10.1056/NEJMoa1602412. Epub 2016 Mar 4. PMID 26943629
- [Derived] Lebov JF, Nason M, Stolka KB, Ximenes R, Mussi-Pinhata MM, Moye J, Zorrilla CD, Velez Vega CM, Cordero JF, Scalabrin DMF, Ko AI, Moreira MEL, Galvao LA, Britt W, Marques ETA, Balmaseda A, Harris E, Arias JF, Schultz-Cherry S, Garces AL, Krebs NF, Ochoa TJ, Ugarte-Gil CA, Fogleman E, Gabriel E, Welton M, Irizarry CM, de Moura Negrini SB, Coutinho CM, de Barros Miranda-Filho D, Montarroyos UR, Cordeiro MT, Gajewski A, Osorio JE, Figueroa L. Zika in Infants and Pregnancy (ZIP) study: results from a prospective international cohort study of prenatal Zika virus infection and adverse fetal and infant outcomes. BMC Pregnancy Childbirth. 2025 Aug 30;25(1):903. doi: 10.1186/s12884-025-07774-y. PMID 40885911
- [Derived] Lebov JF, Arias JF, Balmaseda A, Britt W, Cordero JF, Galvao LA, Garces AL, Hambidge KM, Harris E, Ko A, Krebs N, Marques ETA, Martinez AM, McClure E, Miranda-Filho DB, Moreira MEL, Mussi-Pinhata MM, Ochoa TJ, Osorio JE, Scalabrin DMF, Schultz-Cherry S, Seage GR 3rd, Stolka K, Ugarte-Gil CA, Vega CMV, Welton M, Ximenes R, Zorrilla C. International prospective observational cohort study of Zika in infants and pregnancy (ZIP study): study protocol. BMC Pregnancy Childbirth. 2019 Aug 7;19(1):282. doi: 10.1186/s12884-019-2430-4. PMID 31391005